CLINICAL TRIAL: NCT04688450
Title: Live User Acceptance Testing of a Decision Support System to Optimize Blood Pressure Management During Critical Care
Brief Title: BP Management System User Acceptance Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Tomas Reisner (Other)
Collaborators: Nihon Kohden (Industry)
Responsible Party: Sponsor-Investigator, Andrew Tomas Reisner, Attending Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019P000837
Record Dates: First submitted 2020-12-02; First posted 2020-12-30 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hypotension and Shock
Keywords: vasopressor; arterial blood pressure; clinical decision support system
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Intervention Model Description: This is a single arm feasibility study
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention group (Experimental): The investigational system will be evaluated for safety and user acceptance in 20 patient-subjects and associated nurse-subjects
  Interventions: Device: VIGORIS Blood Pressure Management Clinical Decision Support System

INTERVENTIONS:
Device: VIGORIS Blood Pressure Management Clinical Decision Support System — Software system to optimize tight blood pressure management during vasopressor infusion

SUMMARY:
This is a feasibility study for an investigational clinical decision support system ("the System") intended to optimize the management of blood pressure (BP) for patients during vasopressor infusion. The investigational outcomes are the perceptions of the nurse-subjects who are managing the BP of the patient-subjects; the operational performance of the System; and any technical failures of the software during real-time operation.

DETAILED DESCRIPTION:
This is a feasibility study for an investigational clinical decision support system ("the System") intended to optimize the management of blood pressure (BP) for patients during vasopressor infusion. Enrollment is planned of a convenience sample of 20 individual patient-subjects and also the 20 nurse-subjects who correspond to the primary nurses managing the patient-subjects. Consent will be obtained by the investigative team from the patient-subject (or close family member or healthcare proxy) and from the nurse-subject. The nurse will receive training in the intended use and important limitations of the System. The System will be deployed to the patient's bedside and the System will be initiated. This intervention will continue for a duration of between 4 to 8 hours. A Technical Observer ("TO") will be present to continually oversee the operation of the System, watching to ensure that there are no observable technical failures. The TO will also watch to see if any early termination conditions are met (specifically any concerns by the clinical staff or the patient or the patient's family; any observed technical operational problems; maximum dose vasopressors or hypoxia despite maximum respiratory support; or unplanned bedside response by the clinical care team) and also will make annotations about the exact time that specific clinical interventions are performed. After the intervention, the nurse-subject will be surveyed. Prior to enrollment of a subsequent subject, additional data analysis -- sufficient to identify or exclude any early stoppage condition -- will be performed on the System's archived electronic data and log files. Any adverse events will be reported to the IRB and the FDA as per FDA and institutional policy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years or older) receiving continuous vasopressor infusion to maintain blood pressure;
* Clinician treating patient estimates future duration of vasopressor infusion likely at least 4 additional hours;
* Provider order has been made that sets lower limit for mean arterial pressure;
* Indwelling arterial catheter has been placed for continuous blood pressure monitoring.

Exclusion Criteria:

* Lack of consent or at the discretion of the patient's primary nurse;
* The discretion of any of the patient's other clinical providers;
* People who do not speak English will be excluded. The rationale is that this protocol involves the bedside deployment of an investigational system plus longitudinal observation. Our mitigation for psychosocial risk involves a continual observer who can monitor for any evidence of subject psychosocial discomfort, which involves the ability to effectively communicate with the subject throughout the duration of the protocol. This therefore excludes patients who do not speak English.
* Patients who are on two simultaneous vasopressors running at maximum doses (per the ICUs own protocols) or who is on one maximum-dose vasopressor and has a contraindication to receiving a second vasopressor (e.g., insufficient vascular access).
* Patients who are hypoxic (SpO2 < 90%) despite maximum inspired oxygen (100% for patients receiving mechanical ventilation, or 10L high-flow in patients who are not candidates for mechanical ventilation).
* Provider order has been made that sets lower limit for SBP (because our system does not have the capability to provide decision-support for an SBP lower limit).
* Enhanced respiratory precautions for COVID.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Reisner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD may be shared if consistent with our institutional policy and approved by Nihon Kohden Innovation Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group
Started | 20
Completed | 18
Not Completed | 2
Not completed — Unable to start software due to serial communication failure | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 67.5 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Nurse-subject Survey Response
Description: Nurse-subject quantitative survey response (yes/no) about any confusion or perceived inaccuracies of the system; perceived risk of patient management error; or perceived distraction that impacted care delivery
Time Frame: Up to 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
Participants
  No confusion or perceived inaccuracies of the system | 13
  Any confusion or perceived inaccuracies of the system but without perceived risk of management error | 4
  Perceived risk of patient management error | 1
  Perceived error or distraction that actually impacted care delivery during investigational protocol | 0
  Did not begin protocol / no survey | 2

2. Primary Outcome: Software Operation (Based on Real-time Observation)
Description: System malfunction (yes/no) observed in real-time by the Technical Observer
Time Frame: Up to 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
Participants
  System malfunction not observed | 18
  System malfunction observed | 0
  Did not begin protocol / no survey | 2

3. Primary Outcome: Data Completeness
Description: Completeness (yes/no) of flowsheet (data archive of the investigational System) without any lapses in input data from the bedside monitor during connectivity; and without lapses in associated BP forecasts.
Time Frame: Up to 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
Participants
  Completeness of flowsheet observed | 18
  Incompleteness of flowsheet observed | 0
  Did not begin protocol / no survey | 2

4. Primary Outcome: Software Operation (Based on Review of Error Logs)
Description: Error-level and critical-level software errors in the runtime log (yes/no)
Time Frame: Up to 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
Participants
  Errors in runtime log not observed | 18
  Errors in runtime log observed | 1
  Did not begin protocol | 1

5. Secondary Outcome: Percentage of Time That the BP Forecast is Operative (Outcome 2.1)
Description: Median percentage (%) of time, per patient, during the session when inclusion criteria were otherwise met that the BP forecast was operative (i.e., time intervals when no InOp criteria detected by the System leading to the InOp state)
Time Frame: up to 8 hours
Population: Out of the 20 total patient-subjects, 2 subjects did not begin the protocol which leaves n=18 for the analysis population.
Measure: Median (Inter-Quartile Range); unit: Percentage of time
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Percentage of time | 89.3 [86.0 to 92.9]

6. Secondary Outcome: Accuracy of the MAP Forecast (Outcome 2.2)
Description: Accuracy of the future 20 min median MAP forecast (average error between the MAP forecast and the future 20 min median MAP; for purposes of computing future 20 min median MAP, MAP < 10 mmHg and MAP > 250 mmHg is treated as a missing number) over time intervals during the session when inclusion criteria were otherwise met; the BP forecast was operative; and the analysis window criteria were met [at least 19 minutes remaining to the end of the record from the time of the forecast; and the analysis window has no more than 9 min of non-physiological MAP data (non-physiological MAP criteria are MAP < 10mmHg or MAP > 250mmHg or 'NaN')].
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
mmHg | 0.2 [-9.3 to 9.7]

7. Secondary Outcome: Percentage of Time That the True Future 20 Min Median MAP Falls Within the Forecast Cone (Outcome 2.3)
Description: Median percentage (%) of time, per patient, that the true future 20 min median MAP falls within the computed forecast cone over time intervals during the session when inclusion criteria were otherwise met; the BP forecast was operative; and the analysis window criteria were met [at least 19 minutes remaining to the end of the record from the time of the forecast; and the analysis window has no more than 9 min of non-physiological MAP data (non-physiological MAP criteria are MAP < 10mmHg or MAP > 250mmHg or 'NaN')]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage of time
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Percentage of time | 99.4 [97.0 to 100.0]

8. Secondary Outcome: SHE Incidence (Outcome 3.1)
Description: SHE incidence per 24 hrs [Sustained hypotensive event "SHE" is any interval commencing upon MAP < goal & 20-min future median MAP is also < goal; terminating upon time point when MAP >= goal and & 20-min future median MAP >= goal; SHEs occurring sequentially within 10 min are merged; any remaining SHEs not persisting at least 10 min are excluded]. [Clarification: We are reporting the mean "events per patient-day" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Events per patient-day (24 hours)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Events per patient-day (24 hours) | 4.2

9. Secondary Outcome: Percentage of Total SHEs Predicted by {Index > 35%} Prior to Earliest Hypotension (Outcome 3.2.1)
Description: Percentage (%) of total SHEs predicted by an SHE-contiguous notification event (i.e., Index > 35%) prior to the SHE's earliest hypotension [hypotension is defined as MAP < goal, with the exclusion of MAP < 10 mmHg, which is treated as a missing number]. Notification events are intervals that begin when there is an Index value that meets the notification criteria and terminate when there is an Index value output that does not meet the notification criteria.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total SHE events
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Percentage of total SHE events | 69.2

10. Secondary Outcome: Advance Warning Times (AWTs) for SHEs Predicted by {Index > 35%} Prior to Earliest Hypotension (Outcome 3.2.2)
Description: AWTs (median) for SHEs predicted by an SHE-contiguous notification event (i.e., Index > 35%) prior to the SHE's earliest hypotension [i.e., MAP < goal]. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Minutes | 6.8 [1.5 to 55.3]

11. Secondary Outcome: Percentage of Total SHEs Predicted by {Index > User's Index Threshold Setting} Prior to Earliest Hypotension (Outcome 3.2.3)
Description: Percentage (%) of total SHEs predicted by an SHE-contiguous notification event (i.e., Index > user's Index threshold setting) prior to the SHE's earliest hypotension [i.e., MAP < goal]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total SHE events
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Percentage of total SHE events | 69.2

12. Secondary Outcome: AWTs for SHEs Predicted by {Index > User's Index Threshold Setting} Prior to Earliest Hypotension (Outcome 3.2.4)
Description: AWTs for SHEs predicted by an SHE-contiguous notification event (i.e., Index > user's Index threshold setting) prior to the SHE's earliest hypotension [i.e., MAP < goal]. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Minutes | 6.8 [1.5 to 55.3]

13. Secondary Outcome: Percentage of Total SHEs Predicted by {Index > 35%} Prior to Continuous Hypotension (Outcome 3.3.1)
Description: Percentage (%) of total SHEs predicted by an SHE-contiguous notification event (i.e., Index > 35%) prior to continuous hypotension [intervals of ≥ 10 minutes of physiological MAP continuously below the hypotension threshold (physiological MAP are samples that do not meet the non-physiological criteria)]. NOTE: excluding SHEs predicted prior to earliest hypotension
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total SHE events
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Percentage of total SHE events | 30.8

14. Secondary Outcome: AWTs for SHEs Predicted by {Index > 35%} Prior to Continuous Hypotension (Outcome 3.3.2)
Description: AWTs for SHEs predicted by an SHE-contiguous notification event (i.e., Index > 35%) prior to continuous hypotension and excluding SHEs predicted prior to earliest hypotension. NOTE: A negative AWT denotes a notification event that occurs chronologically after the onset of the SHE event. For example, an AWT of -3 would mean the first notification event occurred 3 minutes after the onset of the SHE event, although still in advance of continuous hypotension.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Minutes | -2.9 [-3.8 to -1.9]

15. Secondary Outcome: Percentage of Total SHEs Predicted by {Index > User's Index Threshold Setting} Prior to Continuous Hypotension (Outcome 3.3.3)
Description: Percentage (%) of total SHEs predicted by an SHE-contiguous notification event (i.e., Index > user's Index threshold setting) prior to continuous hypotension [intervals of ≥ 10 minutes of physiological MAP continuously below the hypotension threshold (physiological MAP are samples that do not meet the non-physiological criteria)]. NOTE: excluding SHEs predicted prior to earliest hypotension
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total SHE events
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Percentage of total SHE events | 30.8

16. Secondary Outcome: AWTs for SHEs Predicted by {Index > User's Index Threshold Setting} Prior to Continuous Hypotension (Outcome 3.3.4)
Description: AWTs for SHEs predicted by an SHE-contiguous notification event (i.e., Index > user's Index threshold setting) prior to continuous hypotension and excluding SHEs predicted prior to earliest hypotension. NOTE: A negative AWT denotes a notification event that occurs chronologically after the onset of the SHE event. For example, an AWT of -3 would mean the first notification event occurred 3 minutes after the onset of the SHE event, although still in advance of continuous hypotension.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Minutes | -3.8 [-5.0 to -2.4]

17. Secondary Outcome: Percentage of Total SHEs Detected by {Index > 35%} After Continuous Hypotension Onset (Outcome 3.4.1)
Description: Percentage (%) of total SHEs predicted by an SHE-contiguous notification event (i.e., Index > 35%) after onset of continuous hypotension
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total SHE events
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Percentage of total SHE events | 0.0

18. Secondary Outcome: AWTs for SHEs Predicted by {Index > 35%} After Continuous Hypotension Onset (Outcome 3.4.2)
Description: AWTs for SHEs predicted by an SHE-contiguous notification event (i.e., Index > 35%) after onset of continuous hypotension. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Minutes | NA [NA to NA] — There were no SHE events predicted by a SHE-contiguous notification event (i.e., Index > 35%) after onset of continuous hypotension, thus AWT is N/A.

19. Secondary Outcome: Percentage of Total SHEs Detected by {Index > User's Index Threshold Setting} After Continuous Hypotension Onset (Outcome 3.4.3)
Description: Percentage (%) of total SHEs predicted by an SHE-contiguous notification event (i.e., Index > user's Index threshold setting) after onset of continuous hypotension
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total SHE events
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Percentage of total SHE events | 0.0

20. Secondary Outcome: AWTs for SHEs Predicted by {Index > User's Index Threshold Setting} After Continuous Hypotension Onset (Outcome 3.4.4)
Description: AWTs for SHEs predicted by an SHE-contiguous notification event (i.e., Index > user's Index threshold setting) after onset of continuous hypotension. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Minutes | NA [NA to NA] — There were no SHE events predicted by a SHE-contiguous notification event (i.e., Index > user's Index threshold setting) after onset of continuous hypotension, thus AWT is N/A.

21. Secondary Outcome: Percentage of Total SHEs With False Resolutions (Outcome 3.5.1)
Description: Percentage of total SHEs with false resolutions [i.e., MAP >= goal transiently during SHE]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total SHE events
Units Other Than Participants: Sustained hypotensive events (SHE)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Sustained hypotensive events (SHE)) | 13
Percentage of total SHE events | 100.0

22. Secondary Outcome: Percentage of Total SHE False Resolutions Detected by {Index > 35%} (Outcome 3.5.2)
Description: Percentage (%) of total SHE false resolutions with a contiguous notification event where {Index > 35%}
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total false resolutions
Units Other Than Participants: SHE false resolutions
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (SHE false resolutions) | 354
Percentage of total false resolutions | 96.3

23. Secondary Outcome: Percentage of Total SHE False Resolutions Not Detected by {Index > 35%} With InOp State During False Resolution (Outcome 3.5.3)
Description: Percentage of total SHE false resolutions that were not detected by {Index > 35%} and had InOp state occurring during the index false resolution episode
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total false resolutions
Units Other Than Participants: SHE false resolutions
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (SHE false resolutions) | 354
Percentage of total false resolutions | 0.3

24. Secondary Outcome: Percentage of Total SHE False Resolutions Not Detected by {Index > 35%} Without InOp State During False Resolution (Outcome 3.5.4)
Description: Percentage (%) of total SHE false resolutions that were not detected by {Index > 35%} and did not have InOp state occurring during the index false resolution episode
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total false resolutions
Units Other Than Participants: SHE false resolutions
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (SHE false resolutions) | 354
Percentage of total false resolutions | 3.4

25. Secondary Outcome: Percentage of Total SHE False Resolutions Detected by {Index > User's Index Threshold Setting} (Outcome 3.5.5)
Description: Percentage (%) of total SHE false resolutions with a contiguous notification event where {Index > user's Index threshold setting}
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total false resolutions
Units Other Than Participants: SHE false resolutions
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (SHE false resolutions) | 354
Percentage of total false resolutions | 95.2

26. Secondary Outcome: Percentage of Total SHE False Resolutions Not Detected by {Index > User's Index Threshold Setting} With InOp State During False Resolution (Outcome 3.5.6)
Description: Percentage (%) of total SHE false resolutions that were not detected by {Index > user's Index threshold setting} and had InOp state occurring during the index false resolution episode
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total false resolutions
Units Other Than Participants: SHE false resolutions
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (SHE false resolutions) | 354
Percentage of total false resolutions | 0.3

27. Secondary Outcome: Percentage of Total SHE False Resolutions Not Detected by {Index > User's Index Threshold Setting} Without InOp State During False Resolution (Outcome 3.5.7)
Description: Percentage (%) of total SHE false resolutions that were not detected by {Index > user's Index threshold setting} and did not have InOp state occurring during the index false resolution episode
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total false resolutions
Units Other Than Participants: SHE false resolutions
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (SHE false resolutions) | 354
Percentage of total false resolutions | 4.5

28. Secondary Outcome: Incidence of Notification Events {Index > 35%} That Are Contiguous With SHEs (Outcome 3.6.1)
Description: Incidence of notification events {Index > 35%} that are contiguous with SHEs, excluding notification events with onset during an SHE. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 2.3

29. Secondary Outcome: Incidence of Notification Events {Index > User's Index Threshold Setting} That Are Contiguous With SHEs (Outcome 3.6.2)
Description: Incidence of notification events {Index > user's Index threshold setting} that are contiguous with SHEs, excluding notification events with onset during an SHE. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 2.3

30. Secondary Outcome: Incidence of Notification Events {Index > 35%} That Are Sentinel Notifications (Outcome 3.6.3)
Description: Incidence of notification events {Index > 35%} that are sentinel notifications [sentinel notification is a notification event that occurs within 60 min prior to an SHE; recorded dose increase; or during stuttering hypotension (defined in 3.7.1)], excluding notification events with onset during an SHE. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 7.8

31. Secondary Outcome: Incidence of Notification Events {Index > User's Index Threshold Setting} That Are Sentinel Notifications (Outcome 3.6.4)
Description: Incidence of notification events {Index > user's Index threshold setting} that are sentinel notifications, excluding notification events with onset during an SHE. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 7.1

32. Secondary Outcome: Incidence of Notification Events {Index > 35%} That Are False Notifications (Outcome 3.6.5)
Description: Incidence of notification events {Index > 35%} that are false notifications (defined as notification events not contiguous with an SHE and not a sentinel notification, excluding notification events with onset during an SHE. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 10.0

33. Secondary Outcome: Incidence of Notification Events {Index > User's Index Threshold Setting} That Are False Notifications (Outcome 3.6.6)
Description: Incidence of notification events {Index > user's Index threshold setting} that are false notifications. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 10.7

34. Secondary Outcome: Incidence of Notification Events {Index > 35%} Contiguous With an SHE False Resolution (Outcome 3.6.7)
Description: Incidence of notification events {Index > 35%} contiguous with an SHE false resolution. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 3.2

35. Secondary Outcome: Incidence of Notification Events {Index > User's Index Threshold Setting} Contiguous With an SHE False Resolution (Outcome 3.6.8)
Description: Incidence of notification events {Index > user's Index threshold setting} contiguous with an SHE false resolution. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 3.6

36. Secondary Outcome: Incidence of Notification Events {Index > 35%} Contiguous With an SHE True Resolution, Overall (Outcome 3.6.9)
Description: Incidence of notification events {Index > 35%} contiguous with an SHE true resolution. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 3.6

37. Secondary Outcome: Incidence of Notification Events {Index > User's Index Threshold Setting} Contiguous With an SHE True Resolution, Overall (Outcome 3.6.10)
Description: Incidence of notification events {Index > user's Index threshold setting} contiguous with an SHE true resolution. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 3.6

38. Secondary Outcome: Incidence of Notification Events {Index > 35%} Contiguous With an SHE True Resolution, Suppressible (Outcome 3.6.11)
Description: Incidence of notification events {Index > 35%} contiguous with an SHE true resolution after excluding all notification event interval that were within 8 min of a documented clinical intervention. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 0.7

39. Secondary Outcome: Incidence of Notification Events {Index > User's Index Threshold Setting} Contiguous With an SHE True Resolution, Suppressible (Outcome 3.6.12)
Description: Incidence of notification events {Index > user's Index threshold setting} contiguous with an SHE true resolution after excluding all notification event interval that were within 8 min of a documented clinical intervention. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 0.7

40. Secondary Outcome: Incidence of Notification Events {Index > 35%} With Onset During an SHE (Outcome 3.6.13)
Description: Incidence of notification events {Index > 35%} with onset during an SHE. [Clarification: We are reporting the mean "notification events / patient-day (24h)" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 1.3

41. Secondary Outcome: Incidence of Notification Events {Index > User's Index Threshold Setting} With Onset During an SHE (Outcome 3.6.14)
Description: Incidence of notification events {Index > user's Index threshold setting} with onset during an SHE. [Clarification: We are using "notification events / patient-day (24h)" as the Unit of Measure for several reasons. First, different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Notification events / patient-day (24h)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Notification events / patient-day (24h) | 1.3

42. Secondary Outcome: Duration of False Notification Events {Index > 35%} (Outcome 3.6.15)
Description: Median duration of false notification events {Index > 35%}
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Notification events
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Notification events) | 66
Minutes | 3.8 [2.0 to 7.7]

43. Secondary Outcome: Duration of False Notification Events {Index > User's Index Threshold Setting} (Outcome 3.6.16)
Description: Median duration of false notification events {Index > user's Index threshold setting}
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Notification events
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Notification events) | 66
Minutes | 3.8 [2.0 to 8.4]

44. Secondary Outcome: Stuttering Hypotension Incidence (Outcome 3.7.1)
Description: Stuttering hypotension incidence [Stuttering hypotension event commences upon hypotension and with >= 10 min of cumulative hypotension within subsequent 60 min; terminates upon next time point when onset condition is no longer met AND when MAP >= goal; intervals that qualify as an SHE are excluded from stuttering hypotension]. [Clarification: We are reporting the mean "events per patient-day" as the Unit of Measure. Different subjects were observed for different intervals of time, with a maximum 8 hours specified in the protocol. Because subjects were observed for different time intervals, it is helpful to standardize findings as events per unit of time. Standardizing the events to units of time allows for valid inter-subject comparison when subjects have differing observation intervals. Next, events per DAY is a conventional Unit of Measurement that is both valid and easy to interpret, even though subjects were not observed for an entire day.]
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Events per patient-day (24 hours)
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Events per patient-day (24 hours) | 3.2

45. Secondary Outcome: Percentage of Total Stuttering Hypotension Episodes Detected by {Index > 35%} Prior to the Stuttering Hypotension's First Hypotension (Outcome 3.7.2)
Description: Percentage (%) of total stuttering hypotension episodes detected by {Index > 35%} prior to the stuttering hypotension's first hypotension
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total stuttering events
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Percentage of total stuttering events | 40.0

46. Secondary Outcome: AWTs for Stuttering Hypotension Episodes Detected by {Index > 35%} Prior to the Stuttering Hypotension's First Hypotension (Outcome 3.7.3)
Description: AWTs for stuttering hypotension episodes detected by {Index > 35%} prior to the stuttering hypotension's first hypotension. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Minutes | 1.3 [0.7 to 2.0]

47. Secondary Outcome: Percentage of Total Stuttering Hypotension Episodes Detected by {Index > User's Index Threshold Setting} Prior to the Stuttering Hypotension's First Hypotension (Outcome 3.7.4)
Description: Percentage (%) of total stuttering hypotension episodes detected by {Index > user's Index threshold setting} prior to the stuttering hypotension's first hypotension
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total stuttering events
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Percentage of total stuttering events | 40.0

48. Secondary Outcome: AWTs for Stuttering Hypotension Episodes Detected by {Index > User's Index Threshold Setting} Prior to the Stuttering Hypotension's First Hypotension (Outcome 3.7.5)
Description: AWTs for stuttering hypotension episodes detected by {Index > user's Index threshold setting} prior to the stuttering hypotension's first hypotension. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Minutes | 1.3 [0.7 to 2.0]

49. Secondary Outcome: Percentage of Total Stuttering Hypotension Episodes Detected by {Index > 35%} Prior to 10 Cumulative Min of Hypotension (Outcome 3.7.6)
Description: Percentage (%) of total stuttering hypotension episodes detected by {Index > 35%} prior to the occurrence of 10 cumulative minutes of hypotension within that stuttering hypotension episode (excluding episodes detected prior to first hypotension)
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total stuttering events
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Percentage of total stuttering events | 60.0

50. Secondary Outcome: AWTs for Stuttering Hypotension Episodes Detected by {Index > 35%} Prior to 10 Cumulative Min of Hypotension (Outcome 3.7.7)
Description: AWTs for stuttering hypotension episodes detected by {Index > 35%} prior to 10 cumulative min of hypotension. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Minutes | -8.0 [-19.2 to -2.2]

51. Secondary Outcome: Percentage of Total Stuttering Hypotension Episodes Detected by {Index > User's Index Threshold Setting} Prior to 10 Cumulative Min of Hypotension (Outcome 3.7.8)
Description: Percentage (%) of total stuttering hypotension episodes detected by {Index > user's Index threshold setting} prior to the occurrence of 10 cumulative minutes of hypotension within that stuttering hypotension episode (excluding episodes detected prior to first hypotension)
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total stuttering events
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Percentage of total stuttering events | 60.0

52. Secondary Outcome: AWTs for Stuttering Hypotension Episodes Detected by {Index > User's Index Threshold Setting} Prior to 10 Cumulative Min of Hypotension (Outcome 3.7.9)
Description: AWTs for stuttering hypotension episodes detected by {Index > user's Index threshold setting} prior to 10 cumulative min of hypotension. NOTE: A positive AWT denotes a notification event that occurs chronologically in advance of the onset of the SHE event. For example, an AWT of +3 would mean the first notification event occurred 3 minutes before the onset of the SHE event.
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Minutes | -8.0 [-19.2 to -2.2]

53. Secondary Outcome: Percentage of Total Stuttering Hypotension Episodes Not Detected by {Index > 35%} Prior to 10 Cumulative Min of Hypotension (Outcome 3.7.10)
Description: Percentage (%) of total stuttering hypotension episodes not detected by {Index > 35%} prior to the occurrence of 10 cumulative minutes of hypotension within that stuttering hypotension episode
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total stuttering events
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Percentage of total stuttering events | 0.0

54. Secondary Outcome: Percentage of Total Stuttering Hypotension Episodes Not Detected by {Index > User's Index Threshold Setting} Prior to 10 Cumulative Min of Hypotension (Outcome 3.7.11)
Description: Percentage (%) of total stuttering hypotension episodes not detected by {Index > user's Index threshold setting} prior to the occurrence of 10 cumulative minutes of hypotension within that stuttering hypotension episode
Time Frame: Up to 8 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of total stuttering events
Units Other Than Participants: Stuttering hypotension episodes
Arm/Group | Intervention Group
Number analyzed (Participants) | 18
Number analyzed (Stuttering hypotension episodes) | 10
Percentage of total stuttering events | 0.0

ADVERSE EVENTS:
Time Frame: 4-8 hours (duration of investigational protocol)
Description: Adverse events (AEs) were determined systematically by a real-time technical observer; nurse-subject surveys; and the software logs. Expected AEs in a population of ICU patients on vasopressors included all sustained hypotension episodes; tachyarrhythmias (HR > 150 bpm) or bradyarrhythmias (HR < 50 bpm) that persist for more than ten minutes; need for chest compressions or defibrillation; or any unscheduled bedside response by the ICU care team involving more than the patient's primary nurse.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=20)
Multi-clinician response (Cardiac disorders) | 1 (1)
Sustained hypotensive event (Cardiac disorders) | 9 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=20)
Unable to electronically communicate with GE monitor (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT04688450/Prot_SAP_000.pdf